CLINICAL TRIAL: NCT03680183
Title: Clinical Pharmacokinetics of Tyrosine Kinase Inhibitors in Chinese Patients of Hepatitis B
Brief Title: Clinical Pharmacokinetics of TKIs in Chinese Patients of Hepatitis B (HBV)
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Affiliated Cancer Hospital & Institute of Guangzhou Medical University (Other)
Responsible Party: Principal Investigator, Tian-Tian Cheng, Secretary of GCP, Affiliated Cancer Hospital & Institute of Guangzhou Medical University
Other Study IDs: PTKI-HBV-01
Record Dates: First submitted 2018-09-13; First posted 2018-09-21 (Actual); Last update posted 2018-09-28 (Actual); Status verified 2018-09

CONDITIONS: Non Small Cell Lung Cancer; Hepatitis B
Keywords: Tyrosine kinase inhibitors; pharmacokinetics; Hepatitis B
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Hepatitis B | interventions — entecavir; Tablets; bicyclol

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Biospecimen Retention: Samples Without DNA — 5ml of whole blood is collected before and after the anti-HBV treatment to measure the plasma concentration of TKIs
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

GROUPS / COHORTS (2):
- Pre-exposure: Entecavir 1Mg Oral Tablet
  Interventions: Drug: Entecavir 1Mg Oral Tablet
- Post-exposure: Entecavir 1Mg Oral Tablet
  Interventions: Drug: Entecavir 1Mg Oral Tablet

INTERVENTIONS:
Drug: Entecavir 1Mg Oral Tablet — The anti-HBV treatment includes a anti-HBV antibiotics and a drug of protecting liver cells or decrease alanine aminotransferase (ALT) or aspartate transaminase (AST)
  Other Names: Bicyclol Tablets

SUMMARY:
The study will explore the characteristics in clinical pharmacokinetics of gefitinib, erlotinib,afatinib,osimertinib, crizotinib, apatinib, icotinib in Chinese patients of Non-small-cell lung cancer and hepatitis B. The study is self-controlled. The plasma concentration of tyrosine kinase inhibitors will be analyzed before and after system treatment of HBV.

DETAILED DESCRIPTION:
Tyrosine kinase inhibitors (TKIs) are first line treatment for non-small-cell lung cancer patients with mutations in targeted genes. TKIs are metabolized in liver into inactive metabolites before eliminating from body. Liver function might plays a significant role in inter-individual differences of pharmacokinetics of TKIs. Hepatitis B is a disease of high prevalence in south China. The liver function will be compromised if the infection of hepatitis B virus has not been controlled. This study aims to compare the pharmacokinetics of TKIs before and after controlling HBV with standard treatment in Chinese patients of non-small-cell lung cancer.

ELIGIBILITY:
Inclusion Criteria:

* pathological confirmed non-small-cell lung cancer
* with epidermal growth factor receptor (EGFR) or anaplastic lymphoma kinase (ALK) genetic mutation required by different TKIs
* liver function, ALT and/or AST <= 2*upper limit of normal (ULN)
* diagnosed of chronic hepatitis B
* Hepatitis B negative as controlled group
* receiving one type of TKIs
* Age between 18-70

Exclusion Criteria:

* diagnosed of acute/ active hepatitis B
* diagnosed of AIDS
* unable to make decision because of metastasis to central nervous system

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Chinese patients diagnosed of non-small-cell lung cancer. Controlled group are HBV negative and HBV group are diagnosed of chronic hepatitis B. All subjects should be able to make their own decision and sign informed concerned.
Sampling Method: Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2018-05-22 (Actual); Primary Completion 2019-03-01 (Estimated); Study Completion 2021-12-31 (Estimated)

PRIMARY OUTCOMES:
Average plasma concentration of the drugs (TKIs) | one year after recruit
  compare the concentration of TKIs prior to and after anti-HBV treatment

SECONDARY OUTCOMES:
Incidence of adverse reaction caused by TKIs | one year after recruit
  the adverse reaction of TKIs before and after anti-HBV treatment

CONTACTS AND LOCATIONS:
Overall Officials: Shuzhong Cui, MD, Study Director — Affiliated Cancer Hospital & Institute of Guangzhou Medical University
Locations (1):
- Affiliated Cancer Hospital & Institute of Guangzhou Medical University, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: Undecided